CLINICAL TRIAL: NCT04143373
Title: The Effect of Warm Saline Irrigation on the Amount of Bleeding in Impacted Mandibular Third Molar Surgery: a Split-mouth Single-blinded Randomized Controlled Clinical Trial
Brief Title: Effect of Warm Saline Irrigation on Bleeding in Mandibular Third Molar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: TehranUMS thesis #6234
Record Dates: First submitted 2019-10-20; First posted 2019-10-29 (Actual); Results first posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2017-10

CONDITIONS: Surgical Blood Loss; Third Molar
Keywords: Warm Saline
MeSH Terms: conditions — Blood Loss, Surgical

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Warm saline (Experimental): this site was irrigated during impacted mandibular third molar surgery, with normal saline of 37 ± 1 ° C as for the experimental side.
  Interventions: Procedure: warm saline irrigation
- Room temperature saline (No Intervention): this site was irrigated during impacted mandibular third molar surgery, with normal saline of 25 ± 2 ° C as for the control side.

INTERVENTIONS:
Procedure: warm saline irrigation — The objective of this research was to compare the effect of irrigation during impacted mandibular third molar surgery, with normal saline of 25 ± 2 ° C and 37 ± 1 ° C for control and experimental sides, respectively.
  Arms: Warm saline

SUMMARY:
The objective of this research is to compare the effect of irrigation during impacted mandibular third molar surgery, with normal saline of 25 ± 2 ° C and 37 ± 1 ° C for control and experimental sides, respectively.

DETAILED DESCRIPTION:
The objective of this research is to compare the effect of irrigation during impacted mandibular third molar surgery, with normal saline of 25 ± 2 ° C and 37 ± 1 ° C for control and experimental sides, respectively. For this purpose, 40 mandibular impacted third molars will be randomly allocated to two groups and surgically removed with the abovementioned saline temperatures. Finally, the suctioned liquids and duration of the surgeries will be carefully measured and compared between both sides.

ELIGIBILITY:
Inclusion criteria

* Being a candidate for bilateral mandibular third molar surgery
* Both mandibular third molars must have a similar inclination to the second molar
* Both mandibular third molars must have same Pell & Gregory's classification

Exclusion criteria

* Presence of any systemic condition or using any type of medication
* History of allergy to local anesthetic (LA) solutions
* Patients with an active gag reflex
* Pregnant and post-menopause women
* Patients with pericoronitis or any local inflammation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mahboobe Hasheminasab, DMD, Study Director — School of dentistry, Tehran University of Medical Sciences
Locations (1):
- department of oral and maxillofacial surgery, school of dentistry, Tehran university of medical sciences,, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this study, the Enrollment number not equal to the number of participants who Started because this was a split-person design study in which 20 participants enrolled and within each individual, the left or right sides were allocated randomly for receiving these two types of saline.
Units Other Than Participants: third molar teeth
Groups:
- Room Temperature Saline of 25 ± 2 ° C; Warm Saline of 37 ± 1 ° C: In this study, during impacted mandibular third molar surgery, within each individual, one side was irrigated with room temperature saline of 25 ± 2 ° C as for the control side, while the other side of the same individual, was irrigated with normal saline of 37 ± 1 ° C as for the experimental side.
  Within each individual, the left or right sides were allocated randomly for receiving these two types of saline.
Period: Overall Study
Arm/Group | Room Temperature Saline of 25 ± 2 ° C | Warm Saline of 37 ± 1 ° C
Started | 20; 20 third molar teeth | 20; 20 third molar teeth
Completed | 20; 20 third molar teeth | 20; 20 third molar teeth
Not Completed | 0; 0 third molar teeth | 0; 0 third molar teeth

BASELINE CHARACTERISTICS:
Units Other Than Participants: third molar teeth
Groups:
- All Study Participants: In this study, during impacted mandibular third molar surgery, one side was irrigated with room temperature saline of 25 ± 2 ° C as for the control side, while the other side was irrigated with normal saline of 37 ± 1 ° C as for the experimental side.
  The side for each intervention was determined by a table of random numbers.
Arm/Group | All Study Participants
Number analyzed (Participants) | 20
Number analyzed (third molar teeth) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.40 (5.384)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0

OUTCOME MEASURES:

1. Primary Outcome: Amount of Bleeding in Cubic Centimetre
Description: both sides will be irrigated with 200cc of saline and the suctioned liquids will be carefully measured and compared
Time Frame: Intraoperatively, up to 30 minutes
Measure: Mean (Standard Deviation); unit: Cubic Centimeter
Units Other Than Participants: third molar teeth
Arm/Group | Room Temperature Saline of 25 ± 2 ° C | Warm Saline of 37 ± 1 ° C
Number analyzed (Participants) | 20 | 20
Number analyzed (third molar teeth) | 20 | 20
Cubic Centimeter | 11.95 (2.762) | 8.75 (2.593)

2. Secondary Outcome: Duration of the Surgery in Minutes
Description: both sides will be irrigated with 200cc of saline and the duration of the surgeries will be carefully measured and compared between both sides
Time Frame: Intraoperatively, up to 30 minutes
Measure: Mean (Standard Deviation); unit: minutes
Units Other Than Participants: third molar teeth
Arm/Group | Room Temperature Saline of 25 ± 2 ° C | Warm Saline of 37 ± 1 ° C
Number analyzed (Participants) | 20 | 20
Number analyzed (third molar teeth) | 20 | 20
minutes | 14.65 (1.954) | 14.65 (1.725)

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: Since this surgical procedure is considered as minor oral surgery, and all participants were included only if they had no systemic condition, the number of participants at risk for Serious Adverse Events and All-Cause Mortality is considered as zero.
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT04143373/Prot_SAP_000.pdf